CLINICAL TRIAL: NCT03265678
Title: Identification of a Genomic/Transcriptomic Signature for Ageing and Predisposition to Skin Cancer in Normal Sun-exposed Skin
Brief Title: Skin Ageing Signatures and Cancer
Acronym: SASAC
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 11701
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Skin and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm: Registered participants will undergo a clinical assessment to determine whether they have high or low levels of skin ageing. The study will recruit 5 subjects with low levels of skin ageing and 5 subjects with high levels of skin ageing. Recruited patients will undergo skin punch biopsies, blood sampling and collection of lifestyle data.

SUMMARY:
The aim of this study is to identify genetic patterns in normal ageing skin in order to better understand age-related changes.

Data has suggested that skin ageing has a genetic basis and past studies have identified genes that promote skin aging due to sun exposure.

DETAILED DESCRIPTION:
This study will use new tools in an attempt to understand the small changes that take place in skin and may be linked to skin ageing either due to age or the effect of the sun. Some data suggests that these changes may have a genetic basis.

In this study, the doctor will use a clinical scale to assess the participants skin type, the scale will range from 1-5 with 1 being fairer skin types and 5 being darker skin types. The doctors will select 10 female participants who meet the required skin types (1-4), aged between 55 and 65 years who attend clinics for reasons other than skin cancer or other skin diseases. 5 of these patients will have high levels of skin ageing and 5 will have low levels of skin ageing as defined by a set of pre-defined criteria. The criteria will be identified by examining the skin on the participants face and forearm. The study sponsor will collect skin and blood samples from all participants in the high and low skin ageing groups and these will be sent to a specialist laboratory for DNA and RNA analysis (genetic analysis).

The study sponsor hope that this will help us understand the effects of ageing on skin's normal functions but also help us interpret results coming out of other genetic studies in skin cancer. This information will help to better understand the changes linked with the development of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent prior to admission to this study.
2. Female aged between 55 and 65 years.
3. Willing and able to comply with clinical/photographic assessment and laboratory tests

Exclusion Criteria:

1. Previous history of skin cancer, active inflammatory or other skin condition that in the opinion of the investigator may affect the skin ageing assessment.
2. Feverish symptoms which lasted for ≥48 hours prior to study entry.
3. Currently suffering from or having suffered during the last month, with any common systemic disease except arterial hypertension.
4. Received any of the following treatment for more than 6 months during the last two years: hypo or hyperthyroidism treatment, corticoids, non-steroids anti-inflammatory, antihistamines, immunosuppressive treatments, diuretics, antibiotics, anticoagulants, beta blockers.
5. Currently experiencing or having experienced in the last two months prior to study entry problems affecting the skin of the face or forearm for instance acne, eczema, psoriasis, seborroheic dermatitis, herpes zoster.
6. Currently receiving or having received in the last two months prior to study entry any of the following dermatological treatments for more than 8 days: hormone based cream, retinoid based facial cream, > 8% concentration alpha hydroxy acid based cream, topical steroids, antibiotics and antifungals
7. Previous facial aesthetic treatments such as: lifting, chemical peeling, dermabrasion, electrocoagulation, laser, sclerotherapy, reconstructive surgery, botox injection, filler injection.
8. Currently using a hormone based cream that is applied on the forearm for hormonal replacement therapy.
9. Have had a change in skin colour during within one month prior to study entry due to sun exposure
10. Had a session of UV therapy for treatment purposes or in a beauty salon within one month prior to study entry.
11. Use of a self-tanning product

Ages: 55 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants will be approached for the study
Study Population: Potential participants will be identified amongst patients attending outpatient clinics in dermatology, ophthalmology and other general medical specialities for reasons other than skin cancer or inflammatory skin disease. If required, volunteers will also be recruited by advertising from amongst staff within the hospital and Queen Mary University of London. Participants will be identified by the dermatology consultant or research fellow working on this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Recruitment of 10 patients with high or low skin ageing scores and collection of normal sun exposed and non-sun exposed skin and blood for genetic analysis. | 1 Year
  Identify a genomic/transcriptomic molecular signature for skin ageing by correlation of whole genome sequencing and transcriptomic profiles of normal skin and clinically evaluated skin ageing scores

SECONDARY OUTCOMES:
Whole genome sequencing and transcriptomic analysis of normal skin samples | 1 Year
  Comparison of genomic and transcriptomic molecular signature for skin ageing with known genomic and transcriptomic signatures for cSCC

CONTACTS AND LOCATIONS:
Overall Officials: Prof Catherine Harwood, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom